CLINICAL TRIAL: NCT02784028
Title: Phase I Study Assessing Safety of SGM-101, a Fluorochrome-labeled Anti-carcinoembryonic Antigen Monoclonal Antibody for the Detection of Neoplastic Lesions in Patients With Peritoneal Carcinomatosis From CEA Overexpressing Digestive Cancer
Brief Title: Study in Patients With Peritoneal Carcinomatosis From CEA Overexpressing Digestive Cancer
Acronym: FLUOCAR-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICM-URC-2014/35
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2016-05

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Peritoneal Carcinomatosis; SGM-101
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGM-101 (Experimental): 6 dose levels of SGM-101 (5mg/patient, 7.5mg/patient, 10 mg/patient, 12.5mg/patient , 15 mg/patient - 24 h prior surgery and 15 mg/patient - 48h prior surgery
  Interventions: Other: SGM-101

INTERVENTIONS:
Other: SGM-101 — Administration of SGM-101 prior surgery

SUMMARY:
The digestive cancer is the second cause of death worldwide. The presence of peritoneal carcinomatosis is common in the evolution of this type of cancer, as well as increased levels of ACE. This peritoneal carcinomatosis is often underestimated, this being due to low sensitivity detection means.

In recent years, it has been shown that peritoneal carcinomatosis surgery as complete as possible associated with an intraperitoneal chemotherapy gave better results but still failures associated with the presence of microscopic residual tumors.

The use of SGM -101 (developped by SURGIMAB SAS) allows surgeons to detect tumor nodules of small size very easily, in real-time, during surgery (shown in animals).

DETAILED DESCRIPTION:
The digestive cancer is the second cause of death worldwide. The presence of peritoneal carcinomatosis is common in the evolution of this type of cancer, as well as increased levels of ACE. This peritoneal carcinomatosis is often underestimated, this being due to low sensitivity detection means.

In recent years, it has been shown that peritoneal carcinomatosis surgery as complete as possible associated with an intraperitoneal chemotherapy gave better results but still failures associated with the presence of microscopic residual tumors.

SGM -101 (developped by SURGIMAB SAS) is a fluorescent antibody that binds to ACE which is overespressed at the surface of tumor cells. The use of this fluorescent molecule allows surgeons to detect tumor nodules of small size very easily, in real-time, during surgery (shown in animals).

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologic proven primary or recurrent digestive adenocarcinoma and eligible for hyperthermic intraperitoneal chemoperfusion (HIPEC) procedure,
2. Evidence of peritoneal carcinomatosis, presume resectable, assessed by imaging (CT scan (Computed Tomography Scanner) and / or MRI (Magnetic Resonance Imaging)) or during a previous abdominal surgery,,
3. CEA positivity by immunohistochemistry on specimen of primary tumor or recurrence lesion, or circulating plasma CEA ≥ 2 times the upper limit of normal range (ULN),
4. ECOG (Eastern Cooperative Oncology group) < 1
5. Life expectancy of at least three months,
6. AST (Aspartate AminoTransferase), ALT (Alanine AminoTransferase) and Alkaline Phosphatase levels ≤ 5 times the ULN,
7. Total bilirubin ≤ 1.5 times the ULN, Serum creatinine ≤ 1.5 times the ULN, absolute neutrophils counts ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L and hemoglobin ≥ 9 g/dL,(red blood transfusion is allowed if needed),
8. Patients aged over 18 years old,
9. Patients affiliated to a French Social Security System,
10. Signed informed consent (IC) obtained before any study specific procedures.

Exclusion Criteria:

1. ASA (American Society of Anesthesiologists) score ≥ 3,
2. Anticancer therapy (e.g. chemotherapy, radiotherapy, targeted therapy, concomitant systemic immune therapy, or any experimental therapy) within 4 weeks before inclusion,
3. Known serious immune allergic history,
4. Rate of circulating plasma CEA ≥ 300 ng / ml,
5. Other malignancies either currently active or diagnosed in the last 5 years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma.
6. Female patients pregnant or breastfeeding (pregnancy should be ruled by an assay of βhCG plasma within 7 days prior to administration of the conjugate). Patients with reproductive potential and who are sexually active must agree to have at least two methods of contraception for the duration of treatment (2 weeks before and 8 12 weeks after the administration of SGM-101) Male patients, must use an effective method of contraception (condom with spermicidal foam or gel; true abstinence; or vasectomy throughout the study and up to 12 weeks after last SGM-101 administration).
7. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody or patients with untreated serious infections,
8. Any other concurrent and/or uncontrolled medical condition or metabolic dysfunction, that would, in the investigator's judgment contraindicate her participation in the clinical study
9. Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 18 months
  Determination of the recommended phase II dose

CONTACTS AND LOCATIONS:
Overall Officials: Francois Quenet, Principal Investigator — Institut régional du Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No